CLINICAL TRIAL: NCT01732588
Title: Three Way Randomised CrossOver Study in Healthy Subjects to Compare the Relative Bioavailability of Nanoparticulate OZ439 Delivered Via the Enterion™ Capsule to the Proximal Small Bowel With Orally Administered OZ439 as PIB Suspension and Orally Administered Nanoparticulate
Brief Title: A Comparison of the Bioavailability of OZ439 When Delivered Directly to the Small Intestine, or Via the Oral Route
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MMV_OZ439_12_003
Record Dates: First submitted 2012-10-22; First posted 2012-11-26 (Estimated); Results first posted 2015-02-13 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Healthy Volunteers
Keywords: Bioavailability
MeSH Terms: interventions — artefenomel; OOS-A regimen; Regimen B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Regimen A - 120mg OZ439 PIB (Active Comparator): 120mg single dose of OZ439 as powder in bottle (PIB) formulation
  Interventions: Drug: OZ439 120mg PIB
- Regimen B - 120 mg OZ439 IR caplet (Experimental): 120 mg single dose of OZ439 immediate release (IR) caplet formulation containing nanoparticulate, administered directly via the oral route
  Interventions: Drug: 120 mg OZ439 caplet
- Regimen C - 120 mg OZ439 caplet via Enterion capsule (Experimental): 120 mg single dose of OZ439 caplet formulation containing nanoparticulate, administered orally via the Enterion capsule and delivered to the proximal small bowel
  Interventions: Drug: 120mg OZ439 caplet via Enterion capsule

INTERVENTIONS:
Drug: OZ439 120mg PIB — 120mg dose (as free base) of OZ439 as a solution made up from powder in bottle (PIB)
  Other Names: Regimen A
  Arms: Regimen A - 120mg OZ439 PIB
Drug: 120 mg OZ439 caplet — 120 mg (as free base) of OZ439 immediate-release (IR) caplet formulation containing nanoparticulate, administered directly via the oral route
  Other Names: Regimen B
  Arms: Regimen B - 120 mg OZ439 IR caplet
Drug: 120mg OZ439 caplet via Enterion capsule — 120 mg OZ439 (as free base) in an immediate release (IR) caplet formulation containing nanoparticulate,administered orally via the Enterion capsule and delivered directly to the proximal small bowel (PSB)
  Other Names: Regimen C
  Arms: Regimen C - 120 mg OZ439 caplet via Enterion capsule

SUMMARY:
The purpose of this study is to determine the bioavailability of nanoparticulate OZ439 delivered to the proximal small bowel (PSB) via the Enterion™ capsule relative to oral OZ439 suspension (current "powder in bottle" [PIB]) and oral nanoparticulate OZ439.

The study will also characterise the plasma concentration time profile of OZ439 when delivered via Enterion capsule to the PSB in comparison with OZ439 PIB formulation delivered orally and nanoparticulate OZ439 delivered orally Safety and tolerability of OZ439 formulations will be determined following delivery to the PSB and administered orally

DETAILED DESCRIPTION:
Previous clinical studies with OZ439 have shown variable PK and a food effect. One hypothesis is that this may be related to a 'common ion effect' leading to precipitation of the drug as a less soluble hydrochloride salt in the stomach, resulting in variable absorption of the drug. This study is designed to investigate the possibility of improving the PK profile by delivering the drug directly to the PSB, thereby bypassing the stomach. The study will compare a previously dosed PIB formulation with oral delivery of a nanoparticulate as a caplet formulation. The same caplet formulation containing nanoparticulate will be administered to the PSB via the Enterion capsule.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males, or females of non-childbearing potential ie surgically sterilised or post-menopausal
2. Age 18 to 55 years
3. Body mass index of 18 to 30 kg/m2 inclusive
4. Total body weight >50 kg
5. Healthy as determined by pre-study medical history, physical examination (including body temperature) and 12-lead ECG
6. Must have haematology, clinical chemistry and urinalysis results at screening that are within the reference range or ncs
7. Must agree to use an adequate method of contraception
8. Must demonstrate their ability to swallow an empty size 000 capsule
9. Must be willing and able to communicate and participate in the whole study
10. Must provide written informed consent

Exclusion Criteria:

1. Evidence or history of clinically significant oncological, pulmonary, chronic respiratory, hepatic, cardiovascular, haematological, metabolic, neurological, immunological, nephrological, endocrine or psychiatric disease, or current infection
2. Clinically relevant abnormalities in the ECG (12 standard leads) and/or QTcF >450 ms (males) or >470 ms (females)
3. Evidence or history of clinically significant GI disease or surgery (excluding appendectomy or cholecystectomy)
4. Any condition that could possibly affect drug absorption, eg gastrectomy or diarrhoea
5. History of post-antibiotic colitis
6. History of any drug or alcohol abuse in the past 2 years prior to screening
7. Subjects who have a breath carbon monoxide reading of greater than 10 ppm at screening. Subjects who are tobacco users (including smokers and users of snuff, chewing tobacco and other nicotine or nicotine-containing products) must have stopped use within 90 days before screening
8. Receipt of an investigational drug or participation in another clinical research study within the previous 3 months
9. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
10. Subjects who have previously been enrolled in this study
11. Use of any prescription or non-prescription medications, vitamins, herbal supplements or dietary supplements within 14 days prior to the first dose
12. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab)or human immunodeficiency virus (HIV-1 or HIV-2 antibody) results
13. Positive urine drug screen result
14. History of intolerance or hypersensitivity to artemisinins
15. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
16. Presence or history of allergy requiring treatment; hayfever is allowed unless it is active
17. Donation or loss of >400 mL of blood within the previous 3 months
18. Haemoglobin result below the lower limit of the reference range
19. Regular alcohol consumption in males >21 units per week and females >14 units per week
20. Subjects who do not have suitable veins
21. Acute diarrhoea or constipation in the 7 days before the predicted first study day.
22. Presence of non-removable metal objects in the abdomen
23. Radiation exposure exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years
24. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Macintyre, PhD, Study Director — Medicines for Malaria Venture
Locations (1):
- Quotient Clinical, Nottingham, Nottingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Subjects received a single dose of 120 mg OZ439 PIB oral suspension (Regimen A), then 120 mg OZ439 IR caplet (Regimen B); then 120 mg OZ439 caplet formulation containing nanoparticulate delivered to the PSB via Enterion capsule (Regimen C)
- Sequence 2: Subjects received a single dose of 120 mg OZ439 IR caplet (Regimen B); then 120 mg OZ439 caplet formulation containing nanoparticulate delivered to the PSB via Enterion capsule (Regimen C); then 120 mg OZ439 PIB oral suspension (Regimen A).
- Sequence 3: Subjects received a single dose of 120 mg OZ439 caplet formulation containing nanoparticulate delivered to the PSB via Enterion capsule (Regimen C); then 120 mg OZ439 PIB oral suspension (Regimen A); then 120 mg OZ439 IR caplet (Regimen B).
Period: First Intervention (7 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | 4 | 3 | 4
Completed | 4 | 2 | 4
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Second Intervention (7 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | 4 | 2 | 4
Completed | 4 | 2 | 4
Not Completed | 0 | 0 | 0
Period: Third Intervention (7 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | 4 | 2 | 4
Completed | 4 | 2 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: cross over design so each regimen is represented in each sequence once
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 4 | 3 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (12.0) | 35.3 (14.6) | 36.8 (12.3) | 38.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 3 | 2 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United Kingdom | 4 | 3 | 4 | 11
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.50 (3.7) | 24.67 (0.58) | 26.75 (1.89) | 26.09 (2.47)
weight [Mean (Standard Deviation); unit: kg] | 82.53 (13.44) | 68 (8.86) | 80.83 (1.44) | 77.95 (10.58)

OUTCOME MEASURES:

1. Primary Outcome: OZ439 AUC0-∞
Description: Area under the plasma concentration-time curve from zero to infinity (AUC0-∞)
Time Frame: pre dose, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
Population: PK population included all subjects who received at least 1 dose of IMP and who had sufficient plasma concentration data for PK parameter estimation.
  In addition, for Regimen C only subjects in whom the activation was performed successfully at the target site were included for this regimen.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Regimen A - OZ439 120mg PIB: Single dose of 120 mg OZ439 powder in bottle (PIB) oral suspension
- Regimen B - 120 mg OZ439 IR Caplet: Single dose of 120 mg OZ439 Immediate release (IR) caplet formulation containing nanoparticulate
- Regimen C - 120 mg OZ439 Caplet Via Enterion Capsule: Single dose of 120 mg OZ439 caplet formulation containing nanoparticulate delivered to the PSB via Enterion capsule
Arm/Group | Regimen A - OZ439 120mg PIB | Regimen B - 120 mg OZ439 IR Caplet | Regimen C - 120 mg OZ439 Caplet Via Enterion Capsule
Number analyzed (Participants) | 9 | 10 | 9
ng*h/mL | 1230 (46.5) | 907 (46.3) | 398 (99)

2. Primary Outcome: OZ439 Cmax
Description: The maximum observed plasma drug concentrations (Cmax)
Time Frame: pre dose, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Regimen A - OZ439 120mg PIB | Regimen B - 120 mg OZ439 IR Caplet | Regimen C - 120 mg OZ439 Caplet Via Enterion Capsule
Number analyzed (Participants) | 9 | 10 | 9
ng/mL | 180 (50.5) | 82.7 (73.5) | 35.4 (98.7)

3. Secondary Outcome: OZ439 Tmax
Description: Time of maximum observed plasma drug concentrations (Tmax)
Time Frame: pre dose, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours post dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Regimen A - OZ439 120mg PIB | Regimen B - 120 mg OZ439 IR Caplet | Regimen C - 120 mg OZ439 Caplet Via Enterion Capsule
Number analyzed (Participants) | 9 | 10 | 9
hours | 2 [2 to 4] | 4 [2 to 6] | 4 [2 to 4]

ADVERSE EVENTS:
Time Frame: Adverse events collected from screening (up to 28 days) to follow up visit, ie up to 12 days after last OZ439 administration.
Description: The safety population was to include all subjects who have received at least 1 dose of IMP (ie, 11 subjects). In Sequence 2, one subject dropped out after the first intervention (Regimen B) and did not receive regimen A and C. Therefore the safety population for both regimens A and C includes 10 healthy subjects.
Groups:
- Regimen A - 120mg OZ439 PIB: Single oral dose of 120 mg OZ439 as powder in bottle (PIB) formulation.
- Regimen B - 120 mg OZ439 IR Caplet: Single oral dose of 120 mg OZ439 Immediate release (IR) caplet formulation containing nanoparticulate
- Regimen C - 120 mg OZ439 Caplet Via Enterion Capsule: Single dose of 120 mg OZ439 caplet formulation containing nanoparticulate administered orally via the Enterion capsule
Arm/Group | Regimen A - 120mg OZ439 PIB | Regimen B - 120 mg OZ439 IR Caplet | Regimen C - 120 mg OZ439 Caplet Via Enterion Capsule
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 2/11 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A - 120mg OZ439 PIB (N=10) | Regimen B - 120 mg OZ439 IR Caplet (N=11) | Regimen C - 120 mg OZ439 Caplet Via Enterion Capsule (N=10)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
increased alanine aminotransferase (Investigations) | 1 (1) | 0 (0) | 0 (0)
increased aspartate aminotransferase (Investigations) | 1 (1) | 0 (0) | 0 (0)
abnormal electrocardiogram (Investigations) | 0 (0) | 1 (1) | 0 (0)
abnormal urine analysis (Investigations) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less